CLINICAL TRIAL: NCT06112769
Title: A Correlation Study of Internal Jugular Vein Variability Under Deep Inhalation and Propofol-induced Hypotension
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, Principal investigator, Affiliated Hospital of Jiaxing University
Other Study IDs: 2023-KY-603
Record Dates: First submitted 2023-10-29; First posted 2023-11-01 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hemodynamic
Keywords: Internal jugular vein; propofol; hypotension; hemodynamic
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The correlation between internal jugular vein variability during deep inhalation and the decrease in blood pressure during propofol induction.

DETAILED DESCRIPTION:
1. Ultrasound records at least one quiet breathing cycle and one deep inhalation cycle to calculate IJVV
2. Propofol was infused target-controlled at 4 μg/ml, and changes in arterial blood pressure within 3 minutes of propofol induction were observed.
3. Aim to conduct a prospective observational study to evaluate the correlation between internal jugular vein variability during deep inhalation and the decrease in blood pressure during propofol induction.

ELIGIBILITY:
Inclusion Criteria:

* age over 60 years
* American Society of Anesthesiology (ASA) status Ⅱ-Ⅲ
* Surgery with radial artery puncture
* Propofol induction

Exclusion Criteria:

* BMI≥30kg/m2
* People with short necks;
* Previous hypotension (systolic blood pressure <90mmHg or mean arterial pressure <65mmHg)
* Previous poorly controlled hypertension
* Cardiac insufficiency , EF value<50%
* Upper limb deep vein thrombosis
* History of radiotherapy or neck surgery
* Inability to maintain a supine position for necessary measurements
* Mechanical ventilation status or inability to take deep breaths patients
* gastrointestinal surgery
* patients allergic to propofol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing intravenous general anesthesia surgery at Jiaxing First Hospital
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-10-29 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
IJVV during deep inhalation | 1 year
  IJVV (%) = (diamax - diamin)/[(diamax + diamin)/2] × 100

CONTACTS AND LOCATIONS:
Overall Officials: Qinghe Zhou, Principal Investigator — Affiliated Hospital of Jiaxing University
Locations (1):
- Affiliated Hospital of Jiaxing University, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei XL, Xi YZ, Xie L, Li ZP, Tang HL, Zhou QH. Effects of liquid resuscitation guided by internal jugular vein variability during deep inhalation on preventing propofol-induced hypotension in elderly patients. BMC Anesthesiol. 2025 Jul 17;25(1):350. doi: 10.1186/s12871-025-03227-3. PMID 40676549